CLINICAL TRIAL: NCT00279123
Title: Effects of 2 Different Doses of Pantoprazole on Gastric pH and Recurrent Bleeding in Patients Who Bled From Peptic Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kwong Wah Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPI Trial
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2006-01-19 (Estimated); Status verified 2006-01

CONDITIONS: Peptic Ulcer Hemorrhage
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

INTERVENTIONS:
Drug: pantoprazole infusion
Drug: pantoprazole bolus
Drug: no treatment

SUMMARY:
Endoscopic treatment of bleeding peptic ulcers is effective to prevent rebleeding. Adjuvant medical treatment to increase gastric pH may further decrease rebleeding. Recent studies on potent acid suppression by proton pump inhibitors (PPI) demonstrated the efficacy in preventing rebleeding. Lau demonstrated that high dose intravenous infusion of omeprazole decreased rebleeding in peptic ulcers with stigmata of recent hemorrhage.

There is little data regarding the effect of pantoprazole on bleeding peptic ulcers. Furthermore, the optimal dose of PPI is unknown. Few studies have included measurement of gastric pH in addition to clinical outcome.

This study compares the effect of two doses of intravenous pantoprazole with no acid suppression in bleeding peptic ulcers after endoscopic therapy. In addition to the usual clinical endpoints, gastric pH is monitored to study the relation of pH elevation and the clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting with upper gastrointestinal bleeding with upper endoscopy showing a bleeding peptic ulcer with major stigmata of haemorrhage and after successful endoscopic haemostasis.

Exclusion Criteria:

* previous gastrectomy and vagotomy
* patient taking warfarin
* intake of anti-secretory drugs in the previous 48 hours

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-01

PRIMARY OUTCOMES:
Rebleeding rate within 30 days after endoscopic therapy

SECONDARY OUTCOMES:
Transfusion requirement
duration of hospital stay
need for operative intervention
mortality rate
gastric pH
side effects of pantoprazole

CONTACTS AND LOCATIONS:
Overall Officials: Wai-ka Hung, MBBS, Principal Investigator — Department of Surgery, Kowng Wah Hospital
Locations (1):
- Department of Surgery, Kwong Wah Hospital, Hong Kong, China